CLINICAL TRIAL: NCT00980356
Title: Vildagliptin in New Onset Diabetes After Transplantation - A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Vildagliptin in New Onset Diabetes After Transplantation
Acronym: VINODAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marcus Saemann, Prof. Dr. Marcus Säemann, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT: 2009-14405-14; EK645/2009
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Kidney transplantation; New onset diabetes mellitus after transplantation
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin, 50 mg, peroral (Active Comparator)
  Interventions: Drug: Vildagliptin
- Placebo pill (Placebo Comparator)

INTERVENTIONS:
Drug: Vildagliptin — Patients receive once daily 50 mg Vildagliptin
  Arms: Vildagliptin, 50 mg, peroral

SUMMARY:
The purpose of this study is to determine whether monotherapy with Vildagliptin improve glycemic control in kidney transplanted patients with newly diagnosed New Onset Diabetes after Transplantation (NODAT).

DETAILED DESCRIPTION:
Development of new onset diabetes mellitus after transplantation (NODAT) also called post-transplant diabetes mellitus (PTDM) increases the risk of cardiovascular disease and poor short term clinical outcomes. There is currently no doubt about the fact that NODAT is a condition that needs medical attention and treatment. Although most centers follow treatment regimens for DM type II prospective data about their effectiveness in NODAT are lacking. Little information exists in kidney transplantation regarding conventional glucose-lowering therapies, either oral hypoglycemic agents or traditional insulin regimens. The Aim of this study was to evaluate whether a monotherapy with Vildagliptin improve glycemic control and to assess the safety in kidney transplanted patients with newly diagnosed NODAT.

ELIGIBILITY:
Inclusion Criteria:

• Newly diagnosed NODAT defined by pathologic OGTT (2h, 75mg glucose): glucose ≥ 200mg/dl

* renal transplantation (deceased or living donor) and treatment with the standard immunosuppression at our center, consisting of triple therapy with tacrolimus or cyclosporine A, mycophenolate mofetil or azathioprine, and prednisone.
* stable graft function for more than 6 months post transplant.
* informed consent of the patient

Exclusion Criteria:

* patients with prior history of type 1 or type 2 diabetes
* body mass index (BMI) > 40
* pregnancy
* severe renal impairment (GFR < 30 mL/min./1.73 m2)
* severe liver impairment
* severe blood glucose elevation with the need for therapy with insulin or HbA1c >8.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess whether monotherapy with Vildagliptin improve glycemic control in kidney transplanted patients with newly diagnosed NODAT as judged in OGTT 3 months after treatment start compared to placebo. | 3 months

SECONDARY OUTCOMES:
To assess differences in the change in HbA1c and fasting plasma glucose after 3 months after treatment start and to assess the safety and efficacy of Vildagliptin in renal transplanted patients. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcus D Säemann, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882
- [Derived] Haidinger M, Werzowa J, Hecking M, Antlanger M, Stemer G, Pleiner J, Kopecky C, Kovarik JJ, Doller D, Pacini G, Saemann MD. Efficacy and safety of vildagliptin in new-onset diabetes after kidney transplantation--a randomized, double-blind, placebo-controlled trial. Am J Transplant. 2014 Jan;14(1):115-23. doi: 10.1111/ajt.12518. Epub 2013 Nov 26. PMID 24279801
- [Derived] Haidinger M, Werzowa J, Voigt HC, Pleiner J, Stemer G, Hecking M, Doller D, Horl WH, Weichhart T, Saemann MD. A randomized, placebo-controlled, double-blind, prospective trial to evaluate the effect of vildagliptin in new-onset diabetes mellitus after kidney transplantation. Trials. 2010 Oct 6;11:91. doi: 10.1186/1745-6215-11-91. PMID 20925938